CLINICAL TRIAL: NCT00548015
Title: HELPING HANDS: a Comparison of Short- and Long Term Effects of Alternative Strategies for Promoting Hand Hygiene in Hospital Nurses.
Brief Title: Helping Hands: Promoting Hand Hygiene in Hospital Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Prof. Theo van Achterberg PhD, RN, IQ healthcare Radboud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG000279; ZonMw 945-17-101
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2007-10

CONDITIONS: Handwashing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- State of the Art strategy (Active Comparator): education, reminders, performance feedback,
  Interventions: Behavioral: state-of-the art strategy and extented strategy
- extended strategy (Experimental): state-of-the art and coaching ward manager,modeling of informal leaders, norm and target setting
  Interventions: Behavioral: state-of-the art strategy and extented strategy

INTERVENTIONS:
Behavioral: state-of-the art strategy and extented strategy — state-of-the art: education, reminders, performance feedback, extented:state-of-the art and coaching ward manager,modeling of informal leaders, norm and target setting

SUMMARY:
Hand hygiene prescriptions are the most important measure in the prevention of hospital acquired infections. Yet compliance rates are generally below 50% of all opportunities for hand hygiene adherence. This study will test the short- and long term effects of two strategies for promoting hand hygiene in hospital nurses

ELIGIBILITY:
Inclusion Criteria:

* Hand hygiene opportunities at the point of patient care

Exclusion Criteria:

* Hand hygiene opportunities not concerning patient care like personal hygiene

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of adherence of opportunities for hand hygiene | march 2008, october 2008, may 2009, november 2009

SECONDARY OUTCOMES:
Team climate, Cost effectiveness | december 2008, june 2009

CONTACTS AND LOCATIONS:
Overall Officials: Theo van Achterberg, PhD RN, Study Chair — Centre for Quality of Care Research
Locations (3):
- Netherlands (3):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud University Nijmegen Medical Centre, PObox 9101, Nijmegen
  - Elisabeth Ziekenhuis, Tilburg

REFERENCES:
- [Derived] Huis A, Holleman G, van Achterberg T, Grol R, Schoonhoven L, Hulscher M. Explaining the effects of two different strategies for promoting hand hygiene in hospital nurses: a process evaluation alongside a cluster randomised controlled trial. Implement Sci. 2013 Apr 8;8:41. doi: 10.1186/1748-5908-8-41. PMID 23566429
- [Derived] Huis A, Hulscher M, Adang E, Grol R, van Achterberg T, Schoonhoven L. Cost-effectiveness of a team and leaders-directed strategy to improve nurses' adherence to hand hygiene guidelines: a cluster randomised trial. Int J Nurs Stud. 2013 Apr;50(4):518-26. doi: 10.1016/j.ijnurstu.2012.11.016. Epub 2012 Dec 13. PMID 23245456
- [Derived] Huis A, Schoonhoven L, Grol R, Donders R, Hulscher M, van Achterberg T. Impact of a team and leaders-directed strategy to improve nurses' adherence to hand hygiene guidelines: a cluster randomised trial. Int J Nurs Stud. 2013 Apr;50(4):464-74. doi: 10.1016/j.ijnurstu.2012.08.004. Epub 2012 Aug 28. PMID 22939048
- [Derived] Huis A, Schoonhoven L, Grol R, Borm G, Adang E, Hulscher M, van Achterberg T. Helping hands: a cluster randomised trial to evaluate the effectiveness of two different strategies for promoting hand hygiene in hospital nurses. Implement Sci. 2011 Sep 3;6:101. doi: 10.1186/1748-5908-6-101. PMID 21888660